CLINICAL TRIAL: NCT05152784
Title: Trial of Rapid Activation MaPping Using a nOveL Catheter and Integrated Non-invasivE Imaging in Ventricular Tachycardia
Brief Title: The TRAMPOLINE VT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 293735
Record Dates: First submitted 2021-11-24; First posted 2021-12-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Tachycardia
Keywords: Octaray
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Propensity-matched cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Octaray catheter (Experimental): VT ablation guided by activation mapping using the Octaray catheter and integrated cardiac MRI data.
  Interventions: Device: Octaray catheter
- Standard of care (Active Comparator): Identified retrospectively from registry data: propensity matched-controls undergoing VT ablation guided by substrate-modification alone.
  Interventions: Device: Standard of care

INTERVENTIONS:
Device: Octaray catheter — A high density diagnostic catheter used for substrate and activation mapping.
  Arms: Octaray catheter
Device: Standard of care — VT ablation guided by substrate-mapping alone.
  Arms: Standard of care

SUMMARY:
This non-randomised, prospective trial will examine the feasibility and efficacy of VT ablation guided by activation mapping using the Octaray and Optrell catheters. Annotation algorithms within the CARTO3 electro-anatomical mapping system will be integrated with 3D scar segmentation data from cardiac MRI (ADAS-VT), and extrastimulus voltage mapping will identify sites of interest for focussed activation mapping. The investigators hypothesise that the examination of these data will identify critical target sites for ablation. Intra-procedural diagnostic performance of the Octaray and Optrell catheters will be assessed as the primary outcome, and will be compared with the standard of care. Secondary, clinical outcomes - primarily the need for ICD therapies at 12 months post ablation - will be compared with propensity-matched controls undergoing substrate-based ablation alone. Follow-up MRI scans will review the impact of ablation on the elimination of conduction channels.

ELIGIBILITY:
Inclusion Criteria:

* ICD in situ
* Clinical indication for VT ablation; incessant VT or receiving appropriate ICD therapies for VT despite anti-arrhythmic drugs
* Ischaemic or non-ischaemic heart disease

Exclusion Criteria:

* Valvular heart disease precluding LV access
* Cardiotomy within previous 3 months
* Acute coronary syndrome within 6 weeks
* Dialysis patients
* Coagulopathy/Thrombocytopaenia
* Pregnancy/breastfeeding women
* CMR contraindicated
* Prognosis <12 months
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Correct identification of VT exit site | Intra-procedural
  The site of VT origin suggested by activation mapping will be confirmed by either:
  i) Termination with ablation at this site ii) Entrainment of the tachycardia at this site (concealed fusion with PPI-TCL <30ms and equivalent stimulus-QRS interval to EGM-QRS (30-70% TCL) interval) iii) Pace-mapping (average correlation coefficient >90%)
Completeness of diastolic pathway recording | Intra-procedural
  The VT diastolic interval will be divided into temporal segments:
  i) First third: VT entrance ii) Middle third: VT isthmus iii) Final third: VT exit
  Completeness of diastolic pathway recording will be assessed according to the number of segments in which electrical activity is recorded

SECONDARY OUTCOMES:
Requirement for ICD therapies at 1 year | 12 months following VT ablation
  ICD devices will be interrogated at 3 and 12 months post ablation, or according to clinical need, and the requirement for appropriate anti-tachycardia pacing (ATP) or defibrillation recorded
VT burden | 12 months following VT ablation
  ICD devices will be interrogated at 3 and 12 months post ablation, or according to clinical need, and the number and duration of recorded VT episodes noted
Symptoms related to arrhythmia | 12 months following VT ablation
  The Arrhythmia-specific questionnaire in Tachycardia and Arrhythmia (ASTA) will be completed both before and 12 months following ablation to assess for quantitative change in arrhythmia-related symptomatology
Morphological changes on serial cardiac MRIs | 3 months following VT ablation
  Cardiac MRI (CMR) will be performed before and 3 months post ablation. Changes in functional, volumetric and scar-related data will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- St. Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No